CLINICAL TRIAL: NCT05667935
Title: Shanghai Cognitive Impairment Study of the Elderly Population: SheMountain Cohort
Brief Title: Cognitive Impairment Cohort Study of the Elderly Population in SheMountain
Acronym: SheMountain
Status: Not yet recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SheMountain-01
Record Dates: First submitted 2022-12-13; First posted 2022-12-29 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Alzheimer Disease; Dementia; Neurodegenerative Diseases; Cognitive Impairment; Mild Cognitive Impairment
Keywords: Alzheimer disease; Mild cognitive impairment; cohort; Disease Progression
MeSH Terms: conditions — Alzheimer Disease; Dementia; Neurodegenerative Diseases; Cognitive Dysfunction; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood, morning urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a prospective observational study, which involves a cohort of 2000 all-sex and all-ethnic people aged 60 years and above with permanent residence in Tianma area, SheMountain Town, Songjiang District (suburban area), Shanghai. Demographic information, neuropsychiatric scale, peripheral blood, APOE genotype, brain MRI, speech information, AV45-PET, FDG-PET, Tau-PET, GLP-1R PET, and cholinergic receptor probe (ASEM) PET were collected and analyzed. Follow-up visits were performed twice a year for 4 visits, and neuropsychiatric scales and biological samples were collected at each follow-up visit to construct a diagnostic model for patients with mild cognitive impairment, or Alzheimer's disease, as well as a predictive model for the progression of cognitive impairment.

DETAILED DESCRIPTION:
This study is a prospective observational study, which involves a cohort of 2000 all-sex and all-ethnic people aged 60 years and above with permanent residence in Tianma area, SheMountain Town, Songjiang District (suburban area), Shanghai. Demographic information, neuropsychiatric scale, peripheral blood serum Aβ40, Aβ42, p-tau 181, 217, urine proteomic analysis, APOE genotype analysis, brain MRI, and speech information were collected and analyzed. After initial screening 20% of patients with clinically confirmed MCI and AD were randomly selected for AV45-PET, FDG-PET, Tau-PET, GLP-1R PET, and cholinergic receptor probe (ASEM) PET. Follow-up visits were performed twice a year for 4 visits, and neuropsychiatric scales and biological samples were collected at each follow-up visit to construct a diagnostic model for patients with mild cognitive impairment, or Alzheimer's disease, as well as a predictive model for the progression of cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

1. All genders and all ethnic groups aged 60 and above with permanent residence in Tianma area, SheMountain Town, Songjiang District (suburbs), Shanghai.
2. Agree to collect neuropsychiatric scales, biological samples, imaging and other examination information.
3. Agree to participate in this study and sign the informed consent form. And promise to abide by the research procedures, and cooperate with the implementation of the whole process of research

Exclusion Criteria:

1. Suffering from severe mental illness, tumor cachexia, severe liver and kidney dysfunction and other serious physical diseases and unable to cooperate
2. Uncorrectable visual or auditory impairment that hampers the completion of related examination.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population in this study includes permanent residence in SheMountain Town, Songjiang District (suburbs), Shanghai with all genders and all ethnic groups aged 60 and above.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-12-26 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-01-31 (Estimated)

PRIMARY OUTCOMES:
The change of incidence of cognitive impairment | baseline, 2 year, 4 year, 6 year, 8 year
  Number of participants who covert to AD or mild cognitive impairment (MCI) will be recorded to calculate the incidence.

SECONDARY OUTCOMES:
The change of Mini-Mental State Examination (MMSE) | baseline, 2 year, 4 year, 6 year, 8 year
  MMSE is a brief screening instrument used to assess cognitive function (orientation, memory, attention, ability to name objects, follow verbal/written commands, write a sentence, and copy figures) in elderly participants. Total score ranges from 0 to 30; lower score indicates greater disease severity.
The change of Montreal cognitive assessment-Basic (MoCA) | baseline, 2 year, 4 year, 6 year, 8 year
  MoCA is a brief screening instrument used to assess cognitive function (orientation, memory, attention, ability to name objects, follow verbal/written commands, write a sentence, and copy figures) in elderly participants. Total score ranges from 0 to 30; lower score indicates greater disease severity.
The change of Auditory verbal learning test (AVLT) | baseline, 2 year, 4 year, 6 year, 8 year
  AVLT is a screening instrument used to assess the function of memory. The score in long-term memory (N5) ranges from 0 to 12, with lower scores indicating greater disease severity.
The change of Geriatric Depression Scale (GDS) | baseline, 2 year, 4 year, 6 year, 8 year
  GDS is a neuropsychological scale used to assess the level of depression. The total score ranges from 0 to 30, with higher scores indicating greater disease severity.
The change of 36-Item Short Form Survey (SF-36) | baseline, 2 year, 4 year, 6 year, 8 year
  The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. And it consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
The change of MRI neuroimaging | baseline, 2 year, 4 year, 6 year, 8 year
  Evaluation of brain MRI by high-resolution structural T1 imaging, diffusion tensor imaging, and blood oxygenation level dependent (BOLD) imaging.
Positron emission tomography (PET)-CT | baseline
  Including AV45-PET, FDG-PET, Tau-PET, GLP-1R PET, Cholinergic receptor probe (ASEM) PET will be used to detect the amyloid, Tau burden and AD related GLP-1R as well as Cholinergic receptor change.
The change of blood concentration of Phosphorylated Tau, Concentration of Amyloid β (Aβ) | baseline, 2 year, 4 year, 6 year, 8 year
  Blood serum p-tau 181, p-tau 217, Aβ40 and Aβ42at baseline will be tested. The higher blood p-tau is a strong predictor for AD.
The change of Activities of daily living (ADL) | baseline, 2 year, 4 year, 6 year, 8 year
  ADL is a scale used in healthcare to refer to people's daily self-care activities. Eight factors are rated to produce an overall score on a point scale of 0 to 100. The lower the score the more independence in living.
The change of speech information | baseline, 2 year, 4 year, 6 year, 8 year
  Voice data collection, use a voice recorder to collect the patient's description of "stealing biscuit map" language, and save it in SWV format. And use self-developed ASR speech analysis software (China software copyright number: 2016RS164680) for speech analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided